CLINICAL TRIAL: NCT05353595
Title: The Effect of Mealworm Protein Ingestion on Muscle Protein Synthesis Rates During Recovery From Endurance Type Exercise in Vivo in Humans
Brief Title: The Effect of Mealworm Protein Ingestion on Muscle Protein Synthesis After Running Exercise in Humans
Acronym: Centurion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: METC 21-083
Record Dates: First submitted 2022-04-21; First posted 2022-04-29 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Muscle Protein Synthesis
Keywords: Dietary protein; Insect protein; muscle protein synthesis; muscle anabolism; endurance exercise
MeSH Terms: interventions — Insect Proteins

STUDY DESIGN:
Intervention Model Description: randomized, counter-balanced, cross-over design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: protein and placebo are matched for flavour and provided in dark bottle. Independent person is responsible for drink randomization and preparation. Final blood and muscle analyses are performed by research personnel that was unaware of treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insect protein (Experimental): 0.38g insect protein / kg body mass with vanilla flavouring is provided. In the morning the participant is weighed and based on this weight an independent researcher prepares the protein drink.
  Interventions: Dietary Supplement: Insect protein; Behavioral: Running exercise
- placebo (Placebo Comparator): participants receive the same amount of water (based on body weight) with vanilla flavouring. this drink is also prepared by an independent researcher.
  Interventions: Behavioral: Running exercise

INTERVENTIONS:
Dietary Supplement: Insect protein — Insect protein concentrate retrieved from lesser mealworms.
  Arms: insect protein
Behavioral: Running exercise — 40 minutes of running on a treadmill at 70% heart rate corresponding Vo2peak
  Other Names: treadmill running; endurance exercise

SUMMARY:
Rationale: Consumption of sufficient dietary protein is fundamental to skeletal muscle mass maintenance and overall health. Conventional animal-based protein sources such as meat, poultry, fish, eggs, and dairy are considered high-quality sources of dietary protein. However, the production of sufficient amounts of these conventional animal-based proteins to meet future global food demands will be challenging. Consequently, there is a great interest in more sustainable alternatives for these high-quality protein sources. Edible insects have recently been proposed as a high quality source of dietary protein. Insects are produced on a more viable and sustainable commercial scale and, as such, may contribute to ensuring global food security. Insect derived proteins represent a protein source that combines high quality with a (more) sustainable production. Though insect proteins have been suggested as a solution to secure future global dietary protein needs, there little data to support the bioavailability of insect derived proteins and their capacity to stimulate post-exercise muscle protein synthesis rates in vivo in humans.

Objective: To assess the impact of ingesting mealworm derived protein on muscle protein synthesis rates during recovery from aerobic exercise in a group healthy men and women Study design: randomized, counter-balanced, cross-over design Study population: 20 healthy lean (BMI 18.5-30 kg/m2) young males and females (age: 18-35 y inclusive).

Intervention: Subjects will perform running exercise and consume either 0.38 g per kg bodyweight mealworm protein or a non-caloric placebo. In addition, continuous intravenous tracer infusions will be applied, with plasma and muscle samples collected.

Main study parameters/endpoints: The primary outcome will be post-exercise muscle protein synthesis rates following beverage ingestion.

DETAILED DESCRIPTION:
To assess whether volunteers are eligible to participate in this study, we will invite them to the University for a screening visit. At the start of the screening session, the entire experimental trial will be explained and any potential questions will we answered. Thereafter, the volunteers are asked to read, fill out, and sign the informed consent form. After signing the informed consent form, the participants eligibility will be assessed based on the in- and exclusion criteria. To further asses their eligibility, participants will be asked to fill out a medical questionnaire to assess their general health, use of medication, habitual food intake and physical activity. Body mass (with accuracy of 0.1 kg) and height (with accuracy of 0.01 m) will be determined, and body composition assessed via a Dual Energy X-ray Absorptiometry (DEXA) scan. A DEXA scan is a simple, non-invasive procedure. At the beginning of the procedure, subjects will be asked to lie down on a scan table and they need to remain motionless during the measurements. As the scanner moves, a dual energy beam passes through the targeted skeletal muscle section and is measured by a detector. This procedure is repeated until the whole body is scanned and takes approximately 3 minutes.

The screening sessions will take place in the morning and participants are instructed to not have any breakfast in the morning in order to avoid perturbations in the DEXA scan.

In the event of an unexpected medical finding during the screening, subjects will always be notified. If a subject does not want to receive this notification, he/she cannot participate in the study. Then provide the participant with a commercially available snack. Finally, Vo2peak will be determined by an incremental running test to volitional fatigue using a running treadmill (Technogym, Rotterdam). After a 5 minute warm-up at walking speed (5 km/h), speed will be increased (women 8km/h and men 9 km/h) for three minutes. Next, speed will be increased to 11 km/h for women and 12 km/h for men for two minutes. Subsequently, the running speed will remain equal, however, the incline will increase every 2 minutes by 2% until volitional fatigue. O2 uptake and CO2 excretion (Omnical, Maastricht University, The Netherlands), running speed (v), incline (%) and heart rate (Polar Finland) will be recorded at every interval. Ratings of perceived exertion (RPE) will be determined using the Borg scale 6-20 after completion of the test.

After the screening visit, participants will be provided with a 2 day food and activity log , to be filled out during the 2 days prior to Test Day 1. Following Test Day 1, participants will be provided with a 2 day food and activity log, to be filled out during the 2 days prior to Test Day 2.

During these 2 days, participants are allowed to eat and drink the foods they would normally consume, except from alcoholic beverages and protein supplements. Additionally, participants will need to consume a standardized dinner and snack the evening before the experimental trial, no later than 22:00. This standardized dinner is an 'Aviko maaltijdpannetje' and will be purchased at a regular supermarket. As evening snack a 'Mondelice vanille dessert' and a 'Liga Evergreen' will be provided. The expiration date from the manufacturer will be checked. Meanwhile, the meals will be stored in an appropriate freezer at the dietary kitchen in the Metabolic Research Unit Maastricht (MRUM) at the department of Human Biology. The subjects will receive the dinner meal for the evening before Test Day 1 after the screening session and receive the dinner meal to be consumed the evening before Test Day 2 at the end of the first test day.

All participants will be instructed to refrain from any sort of heavy physical exercise for 2 days before the experimental trial and record their activities in the provided activity log. Participants are asked to replicate their food intake and physical activities in the 2 days before Test Day 1 as closely as possible for Test Day 2.

Each subject will participate in 2 experimental trials lasting ~10h. An outline of the study protocol is shown in Figure 3. Subjects will be instructed to report to the university at 7:45 AM in an overnight fasted and rested state, meaning that participants are not allowed to eat and drink (except for water) from 22:00 the night prior to the experimental trial, and that they will be instructed to come to the university by car or public transportation. After the subjects arrive at the University, we will ask them to put on their shorts, determine their body mass, and assign them to a bed. Subjects will rest in a supine position and a Teflon catheter will be inserted in a heated dorsal hand vein and placed in a hot-box (60°C) for arterialized blood sampling. A baseline blood sample (20 mL) will be collected at t= -210min to determine the amino acid enrichment level prior to the intervention. Following basal blood sample collection, a second Teflon catheter will be inserted into an antecubital vein of the contralateral arm for stable isotope infusion with the amino acids 13C6-phenylalanine and D2-tyrosine. At the start of the isotope infusion, the plasma phenylalanine and tyrosine pools will be primed with a single dose of the tracer solution, directly thereafter the continuous tracer infusion will commence.

During the entire experimental test day, the hand with the dorsal hand catheter will be pre-heated for 10 minutes prior to every blood draw in a hot box at 60°C to increase blood flow. This makes it easier to collect blood and prevents nutrient exchange from blood into other tissues. It therefore allows us to collect nutrient-rich (arterialized) blood from a vein. Arterialized blood samples (10mL) will be collected at t = -180, -120, -60, and 0 min to assess plasma tracer enrichments during the tracer infusion in the resting overnight post-absorptive period. After a pre-infusion period of 30 minutes (t = -180), during which the tracer infusion reaches steady state, a first muscle biopsy will be taken from the m. vastus lateralis to determine the background enrichment. At t=-45 min running exercise will be performed (40 minutes at 70% heart rate corresponding Vo2peak). Subsequently, at t= 0 min a second biopsy will be taken from the same leg in order to assess the basal muscle protein synthetic rate. Immediately after the second biopsy, subjects will consume either will ingest a mealworm protein (~0.38 g per kg bodyweight) or a non-caloric placebo beverage. Subjects will be instructed to consume the meal within ~5 min.

Upon drink ingestion, the stopwatch will be reset (t= 0 min), and arterialized blood samples (10 mL) will be collected at t = 30, 60, 90, 120, 180, 240, 300, and 360 min during the post-prandial period to assess plasma amino acid profiles and enrichments. To determine postprandial muscle protein synthesis (MPS), another 2 biopsies will be taken at t = 180 and t = 360 min following meal ingestion from the contra-lateral leg. The muscle biopsy at t = 180 min will allow for calculating peak MPS. It is generally assumed that peak MPS rates are more meaningful in predicting muscle adaptive outcomes than MPS calculated over a longer period. However, the regular time between protein-rich meal/snack moments is usually more than 3 hours and peak muscle protein synthesis rates may appear at different time points depending on the protein source consumed. Thereby, stimulation of muscle protein synthetic rates following protein ingestion can extend beyond this 3h times point. Therefore, taking a muscle biopsy at t = 360 min allows us to obtain physiological relevant information with regard to the duration of the anabolic response to protein intake. Collectively, with the obtained biopsies we can measure muscle protein synthesis in the resting state (-180 - 0 min), the early period following protein ingestion (0 - 180 min), the late period following protein ingestion (180 - 360 min) and the entire postprandial period (0 - 360 min; main outcome).

During each test day, a total of 4 muscle biopsies will be taken through 4 separate incisions, 2 biopsies from the left leg and 2 biopsies from the right leg. In total 13 times blood samples will be taken during each test day, the first sample that will be collected will be 20mL the subsequent samples 10mL, for a total of 140mL. Additionally, gastro-intestinal (GI) symptoms will be assessed at t = -60, 30, and 180 minutes and palatability at t = 15 min by questionnaires (Appendix F1.2).

Each participant will participate in 2 test days (cross-over design). The test days are identical (as described here above) except from the following:

• test drink: mealworm protein drink on one day, a non-caloric placebo on the other day.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 35 y
* BMI 18.5 - 30 kg/m2
* Having given informed consent

Exclusion Criteria:

* Participating in a structured (progressive) exercise program
* Smoking regularly
* Allergy to house dust mites or crustaceans
* Diagnosed GI tract disorders or diseases
* Diagnosed musculoskeletal disorders
* Diagnosed metabolic disorders (e.g. diabetes)
* Cardiovascular disease
* Hypertension (blood pressure above 140/90 mmHg)
* Donated blood 3 months prior to test day
* Pregnant
* Amenorrhea
* Using third generation oral contraceptives
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories).
* Chronic use of gastric acid suppressing medication
* Chronic use of anti-coagulants
* Recent (<1 year) participation in amino acid tracer (L-[ring-13C6]-phenylalanine and L-[3,5-2H2]-tyrosine studies

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis rates | 0-6 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe using plasma as precursor.

SECONDARY OUTCOMES:
Muscle protein synthesis rates | -3- 0 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe
Muscle protein synthesis rates | 0-3 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe
Muscle protein synthesis rates | 3-6 hours
  Muscle protein synthesis rates are calculated using L-ring-13C6-phenylalanine tracer and provided as 1 integrated value over the specified timeframe
Plasma glucose concentrations | 0-6 hours
  Plasma glucose concentrations
Plasma insulin concentrations | 0-6 hours
  Plasma insulin concentrations
Plasma amino acids concentrations | 0-6 hours
  Plasma amino acids concentrations

OTHER OUTCOMES:
Age in year | baseline
Dietary macronutrient intake | 2 days before test days
  assessed by written dietary intake records
Body mass in kg | baseline
  scale
height in m | baseline
  stadiometer
BMI in kg/m^2 | baseline
  calculated form height and body mass
Whole body lean mass in kg | baseline
  dexa
Appendicular lean mass in kg | baseline
  dexa
bodyfat% | baseline
  dexa
VO2max absolute/relative | baseline
  running test

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University Medical Centre+
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No